CLINICAL TRIAL: NCT03228420
Title: A Post-Market, Multicenter, Prospective, Randomized Clinical Trial Comparing 10 kHz Spinal Cord Stimulation (HF10™ Therapy) Combined With Conventional Medical Management to Conventional Medical Management Alone in the Treatment of Chronic, Intractable, Neuropathic Limb Pain
Brief Title: Comparison of 10 kHz SCS Combined With CMM to CMM Alone in the Treatment of Neuropathic Limb Pain
Acronym: SENZA-PDN
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: Nevro Corp (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: CA2016-5
Record Dates: First submitted 2017-07-12; First posted 2017-07-24 (Actual); Results first posted 2021-08-10 (Actual); Last update posted 2021-08-10 (Actual); Status verified 2021-07

CONDITIONS: Painful Diabetic Neuropathy
MeSH Terms: conditions — Diabetic Neuropathies

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: No

ARMS (2):
- HF10 therapy plus CMM (Active Comparator): The addition of HF10 (10kHz SCS) therapy to Conventional Medical Management
  Interventions: Device: Senza HF10 Therapy
- CMM Alone (Other): Conventional Medical Management
  Interventions: Other: CMM

INTERVENTIONS:
Device: Senza HF10 Therapy — Senza 10kHz Spinal Cord Stimulation
  Arms: HF10 therapy plus CMM
Other: CMM — Conventional Medical Management
  Arms: CMM Alone

SUMMARY:
This post-market study is being conducted to document comparative safety, clinical effectiveness, and cost-effectiveness of the addition of HF10™ therapy to CMM compared with CMM alone in subjects with chronic, intractable, neuropathic lower limb pain due to diabetic neuropathy (Painful Diabetic Neuropathy or PDN). This study is a multi-center, prospective, randomized comparison of the two treatments.

ELIGIBILITY:
Inclusion Criteria:

1. Have been clinically diagnosed with painful diabetic neuropathy (PDN) of the lower limbs.
2. Average pain intensity of ≥ 5 out of 10 cm on the VAS in the lower extremities at enrollment.
3. Have stable neurological status.
4. Be on a stable analgesic regimen.
5. Be 22 years of age or older at the time of enrollment.
6. Be an appropriate candidate for the surgical procedures required in this study.
7. Be capable of subjective evaluation, able to read and understand English-written questionnaires, and able to read, understand and sign the written informed consent in English.
8. Be willing and capable of giving informed consent.
9. Be willing and able to comply with study-related requirements, procedures, and scheduled visits.

Exclusion Criteria:

1. Have a diagnosis of a lower limb mononeuropathy, have had a lower limb amputation, or have large (≥3 cm) and/or gangrenous ulcers of the lower limbs.
2. Have a BMI ≥ 40.
3. Currently prescribed a daily opioid dosage > 120 mg morphine equivalents.
4. Have a medical condition or pain in other area(s), not intended to be treated in this study.
5. Have a current diagnosis of a progressive neurological disease such a multiple sclerosis, chronic inflammatory demyelinating polyneuropathy, rapidly progressive arachnoiditis, brain or spinal cord tumor, central deafferentation syndrome, Complex Regional Pain Syndrome, acute herniating disc, severe spinal stenosis and brachial plexus injury.
6. Have a current diagnosis or condition such as a coagulation disorder, bleeding diathesis, platelet dysfunction, low platelet count, severely diminished functional capacity due to underlying cardiac/pulmonary disease, symptomatic uncontrolled hypertension, progressive peripheral vascular disease or uncontrolled diabetes mellitus that presents excess risk for performing the procedure.
7. Have failed prior SCS, dorsal root ganglion (DRG) stimulation, or peripheral nerve stimulation (PNS) trials for chronic intractable pain.
8. Have significant spinal stenosis, objective evidence of epidural scarring and/or any signs or symptoms of myelopathy.
9. Any previous history of surgery on the posterior elements (laminectomy, posterior fusion) resulting in a compromised epidural space.
10. Be benefitting from an interventional procedure and/or surgery to treat lower limb pain.
11. Have an existing drug pump and/or another active implantable device such as a pacemaker.
12. Have a condition currently requiring or likely to require the use of diathermy or MRI that is inconsistent with Senza system guidelines in the Physician's Manual.
13. Have either a metastatic malignant neoplasm or untreated local malignant neoplasm.
14. Have a life expectancy of less than one year.
15. Have a local infection at the anticipated surgical entry site or an active systemic infection.
16. Be pregnant or plan to become pregnant during the study. Women of childbearing potential who are sexually active must use a reliable form of birth control, be surgically sterile, or be at least 2 years post-menopausal.
17. Have within 6 months of enrollment a significant untreated addiction to dependency producing medications, alcohol or illicit drugs.
18. Be concomitantly participating in another clinical study.
19. Be involved in an injury claim under current litigation.
20. Be a recipient of Social Security Disability Insurance (SSDI).
21. Have a pending or approved worker's compensation claim.
22. Have evidence of an active disruptive psychological or psychiatric disorder or other known condition significant enough to impact perception of pain, compliance with intervention and/or ability to evaluate treatment outcome.

Min Age: 22 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 430 (Actual)
Dates: Start 2017-07-20 (Actual); Primary Completion 2020-05-01 (Actual); Study Completion 2022-12-01 (Estimated)

CONTACTS AND LOCATIONS:
Overall Officials: David Caraway, MD, Study Director — Nevro Corp
Locations (4):
- United States (4):
  - Coastal Orthopedics, Bradenton, Florida
  - Georgia Pain Care, Stockbridge, Georgia
  - Duke University Medical Center, Durham, North Carolina
  - Advanced Pain Management, Greenfield, Wisconsin

REFERENCES:
- [Derived] Klonoff DC, Levy BL, Jaasma MJ, Bharara M, Edgar DR, Nasr C, Caraway DL, Petersen EA, Armstrong DG. Treatment of Painful Diabetic Neuropathy with 10 kHz Spinal Cord Stimulation: Long-Term Improvements in Hemoglobin A1c, Weight, and Sleep Accompany Pain Relief for People with Type 2 Diabetes. J Pain Res. 2024 Sep 18;17:3063-3074. doi: 10.2147/JPR.S463383. eCollection 2024. PMID 39308991
- [Derived] Argoff CE, Armstrong DG, Kagan ZB, Jaasma MJ, Bharara M, Bradley K, Caraway DL, Petersen EA; for Investigators. Improvement in Protective Sensation: Clinical Evidence From a Randomized Controlled Trial for Treatment of Painful Diabetic Neuropathy With 10 kHz Spinal Cord Stimulation. J Diabetes Sci Technol. 2025 Jul;19(4):992-998. doi: 10.1177/19322968231222271. Epub 2024 Jan 9. PMID 38193426
- [Derived] Petersen EA, Stauss TG, Scowcroft JA, Jaasma MJ, Brooks ES, Edgar DR, White JL, Sills SM, Amirdelfan K, Guirguis MN, Xu J, Yu C, Nairizi A, Patterson DG, Tsoulfas KC, Creamer MJ, Galan V, Bundschu RH, Mehta ND, Sayed D, Lad SP, DiBenedetto DJ, Sethi KA, Goree JH, Bennett MT, Harrison NJ, Israel AF, Chang P, Wu PW, Argoff CE, Nasr CE, Taylor RS, Caraway DL, Mekhail NA. Long-term efficacy of high-frequency (10 kHz) spinal cord stimulation for the treatment of painful diabetic neuropathy: 24-Month results of a randomized controlled trial. Diabetes Res Clin Pract. 2023 Sep;203:110865. doi: 10.1016/j.diabres.2023.110865. Epub 2023 Aug 1. PMID 37536514
- [Derived] Petersen EA, Stauss TG, Scowcroft JA, Brooks ES, White JL, Sills SM, Amirdelfan K, Guirguis MN, Xu J, Yu C, Nairizi A, Patterson DG, Tsoulfas KC, Creamer MJ, Galan V, Bundschu RH, Mehta ND, Sayed D, Lad SP, DiBenedetto DJ, Sethi KA, Goree JH, Bennett MT, Harrison NJ, Israel AF, Chang P, Wu PW, Argoff CE, Nasr CE, Taylor RS, Caraway DL, Mekhail NA. High-Frequency 10-kHz Spinal Cord Stimulation Improves Health-Related Quality of Life in Patients With Refractory Painful Diabetic Neuropathy: 12-Month Results From a Randomized Controlled Trial. Mayo Clin Proc Innov Qual Outcomes. 2022 Jul 1;6(4):347-360. doi: 10.1016/j.mayocpiqo.2022.05.003. eCollection 2022 Aug. PMID 35814185
- [Derived] Armstrong DG, Grunberger G. Stimulating Results Signal a New Treatment Option for People Living With Painful Diabetic Neuropathy. J Diabetes Sci Technol. 2023 Sep;17(5):1387-1391. doi: 10.1177/19322968221099542. Epub 2022 Jun 30. PMID 35770993
- [Derived] O'Connell NE, Ferraro MC, Gibson W, Rice AS, Vase L, Coyle D, Eccleston C. Implanted spinal neuromodulation interventions for chronic pain in adults. Cochrane Database Syst Rev. 2021 Dec 2;12(12):CD013756. doi: 10.1002/14651858.CD013756.pub2. PMID 34854473
- [Derived] Petersen EA, Stauss TG, Scowcroft JA, Brooks ES, White JL, Sills SM, Amirdelfan K, Guirguis MN, Xu J, Yu C, Nairizi A, Patterson DG, Tsoulfas KC, Creamer MJ, Galan V, Bundschu RH, Mehta ND, Sayed D, Lad SP, DiBenedetto DJ, Sethi KA, Goree JH, Bennett MT, Harrison NJ, Israel AF, Chang P, Wu PW, Argoff CE, Nasr CE, Taylor RS, Caraway DL, Mekhail NA. Durability of High-Frequency 10-kHz Spinal Cord Stimulation for Patients With Painful Diabetic Neuropathy Refractory to Conventional Treatments: 12-Month Results From a Randomized Controlled Trial. Diabetes Care. 2022 Jan 1;45(1):e3-e6. doi: 10.2337/dc21-1813. No abstract available. PMID 34844993
- [Derived] Petersen EA, Stauss TG, Scowcroft JA, Brooks ES, White JL, Sills SM, Amirdelfan K, Guirguis MN, Xu J, Yu C, Nairizi A, Patterson DG, Tsoulfas KC, Creamer MJ, Galan V, Bundschu RH, Paul CA, Mehta ND, Choi H, Sayed D, Lad SP, DiBenedetto DJ, Sethi KA, Goree JH, Bennett MT, Harrison NJ, Israel AF, Chang P, Wu PW, Gekht G, Argoff CE, Nasr CE, Taylor RS, Subbaroyan J, Gliner BE, Caraway DL, Mekhail NA. Effect of High-frequency (10-kHz) Spinal Cord Stimulation in Patients With Painful Diabetic Neuropathy: A Randomized Clinical Trial. JAMA Neurol. 2021 Jun 1;78(6):687-698. doi: 10.1001/jamaneurol.2021.0538. PMID 33818600
- [Derived] Mekhail NA, Argoff CE, Taylor RS, Nasr C, Caraway DL, Gliner BE, Subbaroyan J, Brooks ES. High-frequency spinal cord stimulation at 10 kHz for the treatment of painful diabetic neuropathy: design of a multicenter, randomized controlled trial (SENZA-PDN). Trials. 2020 Jan 15;21(1):87. doi: 10.1186/s13063-019-4007-y. PMID 31941531

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: Participants underwent screening prior to randomization to verify satisfaction of all inclusion/exclusion criteria. Medical records for enrolled participants were evaluated by independent medical monitors for oversight of appropriate patient selection.
Period: Overall Study
Arm/Group | HF10 Therapy Plus CMM | CMM Alone
Started | 113 | 103
Month-1 | 95 | 101
Month-3 | 93 | 98
Completed | 93 | 98
Not Completed | 20 | 5
Not completed — Lost to Follow-up | 5 | 3
Not completed — Withdrawal by Subject | 10 | 0
Not completed — Adverse Event | 5 | 2

BASELINE CHARACTERISTICS:
Population: All randomized patients
Groups:
- Total: Total of all reporting groups
Arm/Group | HF10 Therapy Plus CMM | CMM Alone | Total
Number analyzed (Participants) | 113 | 103 | 216
Age, Continuous [Mean (Standard Deviation); unit: years] | 60.7 (11.4) | 60.8 (9.9) | 60.8 (10.7)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 43 | 37 | 80
  Male | 70 | 66 | 136
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 2 | 0 | 2
  Asian | 1 | 1 | 2
  Native Hawaiian or Other Pacific Islander | 3 | 1 | 4
  Black or African American | 18 | 13 | 31
  White | 87 | 85 | 172
  More than one race | 2 | 3 | 5
  Unknown or Not Reported | 0 | 0 | 0
Lower limb pain visual analog scale (VAS) score [Mean (Standard Deviation); unit: cm] — Participants indicate pain severity by marking on a 10 cm line between 0 (no pain) and 10 (worst pain imaginable)
  cm | 7.5 (1.6) | 7.1 (1.6) | 7.3 (1.6)

OUTCOME MEASURES:

1. Primary Outcome: Composite of Safety and Effectiveness
Description: Difference between treatment groups in responder rates in subjects without a clinically meaningful neurological deficit compared with baseline. Responder is defined as a subject who has at least 50% reduction in lower limb pain from Baseline as measured by a 10 cm Visual Analog Scale (VAS).
Time Frame: 3 months
Population: Intention-to-treat population including all randomized patients whose status could be determined at the 3-month primary assessment, including patients who failed trial SCS and those who withdrew due to an adverse event at any point after the trial SCS phase in the active treatment arm.
Measure: Count of Participants; unit: Participants
Arm/Group | HF10 Therapy Plus CMM | CMM Alone
Number analyzed (Participants) | 95 | 94
Participants | 75 | 5
Statistical Analysis 1: Comparison: HF10 Therapy Plus CMM vs CMM Alone; Test type: Superiority; p < 0.001, Fisher Exact — 2-sided alpha level of 0.05

2. Secondary Outcome: Pain Scores of 3 or Less
Description: Difference between the treatment groups in proportion of subjects with a lower limb pain VAS score ≤ 3 cm.
Time Frame: 3 months
Reporting Status: Not Posted

3. Secondary Outcome: Crossover Rates
Description: Difference between the treatment groups in crossover rates. Subjects who meet pre-specified criteria may elect to crossover to the other treatment arm at 6-month follow-up.
Time Frame: 6 months
Reporting Status: Not Posted

4. Secondary Outcome: Responder Rates
Description: Difference between the treatment groups in responder rates. Responder is defined as a subject who has at least 50% reduction in lower limb pain from Baseline as measured by a 10 cm Visual Analog Scale (VAS).
Time Frame: 6 months
Reporting Status: Not Posted

5. Secondary Outcome: Remitter Rates
Description: Difference between the treatment groups in the proportion of remitters (remission is defined as having a lower limb pain VAS score of ≤ 3.0 cm for at least 6 months).
Time Frame: 6 months
Reporting Status: Not Posted

6. Secondary Outcome: Neurological Assessment
Description: Difference between the treatment groups in the proportion of subjects with overall improvement from baseline in neurological assessment (motor, sensory, reflex).
Time Frame: 3 months
Reporting Status: Not Posted

7. Secondary Outcome: Neurological Assessment
Description: as for outcome 6
Time Frame: 6 months
Reporting Status: Not Posted

8. Secondary Outcome: Health-related Quality of Life
Description: Difference between the treatment groups in changes in health-related quality of life as assessed by the EuroQol Five Dimensions questionnaire (EQ-5D-5L).
Time Frame: 6 months
Reporting Status: Not Posted

9. Secondary Outcome: Hemoglobin A1c
Description: Difference between the treatment groups in the average percentage change from baseline in HbA1c levels.
Time Frame: 6 months
Reporting Status: Not Posted

ADVERSE EVENTS:
Time Frame: 3 months
Arm/Group | HF10 Therapy Plus CMM | CMM Alone
All-Cause Mortality (participants affected / at risk) | 1/113 | 0/103
Serious Adverse Events (participants affected / at risk) | 12/113 | 9/103
Other Adverse Events (participants affected / at risk) | 0/113 | 0/103
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | HF10 Therapy Plus CMM (N=113) | CMM Alone (N=103)
Acute kidney injury (Renal and urinary disorders) | 0 (0) | 1 (1)
Acute myocardial infarction (Cardiac disorders) | 1 (1) | 1 (1)
Diarrhoea (Gastrointestinal disorders) | 0 (0) | 1 (1)
Sepsis (Infections and infestations) | 1 (1) | 1 (1)
Localised infection (Infections and infestations) | 1 (1) | 0 (0)
Extradural haematoma (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Paraplegia (Nervous system disorders) | 1 (1) | 0 (0)
Headache (Nervous system disorders) | 0 (0) | 1 (1)
Nausea (Gastrointestinal disorders) | 0 (0) | 1 (1)
Hypotension (Vascular disorders) | 1 (1) | 0 (0)
Coronary artery disease (Cardiac disorders) | 1 (1) | 0 (0)
Orthostatic hypotension (Vascular disorders) | 1 (1) | 0 (0)
Wound infection staphylococcal (Infections and infestations) | 0 (0) | 1 (1)
Embolic stroke (Nervous system disorders) | 0 (0) | 1 (1)
Encephalopathy (Nervous system disorders) | 0 (0) | 1 (1)
Hypertensive emergency (Vascular disorders) | 0 (0) | 1 (1)
Cervical vertebral fracture (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
Pneumonia (Infections and infestations) | 1 (1) | 1 (1)
Septic shock (Infections and infestations) | 0 (0) | 1 (1)
Staphylococcal infection (Infections and infestations) | 0 (0) | 1 (1)
Acute respiratory failure (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
Chest pain (General disorders) | 1 (1) | 0 (0)
Pyrexia (General disorders) | 1 (1) | 0 (0)
Cholangitis acute (Hepatobiliary disorders) | 1 (1) | 0 (0)
Pancreatic mass (Gastrointestinal disorders) | 1 (1) | 0 (0)
Pancreatitis chronic (Gastrointestinal disorders) | 1 (1) | 0 (0)
Pancreatic disorder (Gastrointestinal disorders) | 0 (0) | 1 (1)
Osteoarthritis (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0)
Cardiac arrest (Cardiac disorders) | 1 (1) | 0 (0)
Wound infection (Infections and infestations) | 1 (1) | 0 (0)
Endocarditis (Infections and infestations) | 0 (0) | 1 (1)
Myocardial infarction (Cardiac disorders) | 0 (0) | 1 (1)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
Initial publication of the results will be a joint, multicenter publication with all PIs and sites contributing data, analyses, and critical review of the manuscript. If no such publication occurs within 12 months of study completion, individual PIs may publish results from their center. PIs will allow sponsor 30 days to review any potential publications or presentations and sponsor can request an additional 60 days if needed.

DOCUMENTS (2):
  • Study Protocol (2019-03-19): https://cdn.clinicaltrials.gov/large-docs/20/NCT03228420/Prot_000.pdf
  • Statistical Analysis Plan (2019-09-15): https://cdn.clinicaltrials.gov/large-docs/20/NCT03228420/SAP_001.pdf